CLINICAL TRIAL: NCT01003769
Title: A Phase I/II Clinical Trial of Lenalidomide in Combination With AT-101 for the Treatment of Relapsed B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: Lenalidomide and AT-101 in Treating Patients With Relapsed B-Cell Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC128A; NCI-2009-01569 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC128A (Other: Mayo Clinic in Florida); P30CA015083 (NIH); 3938 (Other Grant/Funding Number: FDA OOPD); NCT01021345 (obsolete NCT alias)
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide in combination with AT-101) (Experimental): Patients receive lenalidomide PO QD on days 1-21. Beginning in course 2, patients also receive AT-101 PO BID on days 1-3. Treatment repeats every 28 days for up to 11 courses (49-56 days for course 12 or last course of treatment) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Drug: R-(-)-Gossypol Acetic Acid; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; IMiD-1
Drug: R-(-)-Gossypol Acetic Acid — Given PO
  Other Names: (-)-Gossypol Acetic Acid; AT-101
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with R-(-)-gossypol acetic acid and to see how well they work in treating patients with B-cell chronic lymphocytic leukemia (B-CLL) that has returned after a period of improvement (relapsed). Biological therapies, such as lenalidomide, may stimulate the immune system to attack cancer cells. R-(-)-gossypol acetic acid may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and causing the cells to die. Giving lenalidomide with R-(-)-gossypol acetic acid may be an effective treatment for relapsed or refractory B-CLL. - Funding Source - FDA OOPD

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of lenalidomide in combination with AT-101 (R-(-)-gossypol acetic acid). (Phase I) II. To assess the overall response rate of lenalidomide in combination with AT-101. (Phase II)

SECONDARY OBJECTIVES:

I. To assess the overall response rates of lenalidomide in combination with AT-101 at 6 months and 12 months.

II. To evaluate time to progression (TTP) for the combination of lenalidomide + AT-101.

III. To evaluate the safety of this combination in patients with relapsed B-CLL.

TERTIARY OBJECTIVES:

I. To conduct correlative studies for further understanding of the mechanism of antitumor activity of lenalidomide and lenalidomide + AT-101.

OUTLINE: This is a phase I dose-escalation study of lenalidomide followed by a phase II study.

Patients receive lenalidomide orally (PO) once daily (QD) on days 1-21. Beginning in course 3, patients also receive AT-101 PO twice daily (BID) on days 1-3. Treatment repeats every 28 days for up to 11 courses (49-56 days for course 12 or last course of treatment) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Diagnosis of B-CLL, confirmed by flow cytometric analysis and as per the criteria outlined by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL)/Hallek December 2008
* Any prior therapy for B-CLL must have been discontinued >= 28-days prior to registration
* Patients must have absolute lymphocyte counts (ALC) of more than 5,000 cell/mm^3
* During phase I: all patients with relapsed disease will be eligible if they have received at least 1 prior standard CLL therapy and no more than 4 prior therapies (one of which must be a purine analog and/or an alkylating agent)
* During phase II: all patients with relapsed disease will be eligible if they have received a minimum of 1 prior standard therapy and a maximum of 2 prior treatments (one of which must be a purine analog and/or an alkylating agent) for B-CLL and have developed relapse disease

  * Note: patients who have refractory disease (defined as - progressive disease on last treatment, or less than 6 months of clinical response to the last treatment) will not be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at registration
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 30,000/mm^3
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 mg/dL or direct bilirubin =< 1.0 mg/dL for patients with Gilberts syndrome
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2 x ULN or =< 5 x ULN if hepatic disease is present
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL 10-14 days prior to and again within 24 hours before starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure

  * A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Patient must require treatment for symptomatic B-CLL as defined by the by the IWCLL/Hallek, December 2008 criterion or as determined clinically necessary by the treating physician
* Willing to provide blood and baseline bone marrow aspirate samples for correlative research purposes

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Use of any other experimental drug or therapy =< 28 days prior to registration
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Patients with of history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix, unless in complete remission and off therapy for that disease for > 3 years)
* Patient with history of cardiac arrest within the past 6 months
* Patients with history of prior bowel resection, malabsorption syndrome, inflammatory bowel disease, prior bowel obstruction (partial or complete), Crohn disease, or any other disease significantly affecting the gastrointestinal tract
* Prior use of gossypol or AT-101

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher Chanan-Khan, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Roswell Park Cancer Institute, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Lenalidomide in Combination With AT-101): Patients receive 5 mg lenalidomide PO QD on days 1-21. Beginning in course 2, patients also receive 40 mg AT-101 PO BID on days 1-3. Treatment repeats every 28 days for up to 11 courses (49-56 days for course 12 or last course of treatment) in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients registered to Dose Level 1 are included in this analysis.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 61 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: Maximum tolerated dose of lenalidomide when given in combination with AT-101, defined as the dose level below the lowest dose that induces dose limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) (Phase I)
Time Frame: Up to day 28 of course 2
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

2. Primary Outcome: Overall Response Rate (Complete Response [CR], CR With Incomplete Marrow Recovery, Clinical CR, Nodular Partial Response [PR], and PR) (Phase II)
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner.
Time Frame: Up to 2 years
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

3. Secondary Outcome: Incidence of Adverse Events, Graded According to the Grading Scale for Hematologic Adverse Events in CLL Studies (Phase I)
Description: The number and severity of all adverse events (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Time Frame: Up to 2 years
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Toxicity, Defined as Adverse Events Classified as Possibly, Probably, or Definitely Related to Study Treatment, Graded According to the Grading Scale for Hematologic Adverse Events in CLL Studies or Ordinal Common Toxicity Criteria (Phase I)
Description: Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses. Here, we report the number of patients that reported a grade 2 or higher as their worst incidence of toxicity.
Time Frame: Up to 2 years
Population: All patients that were registered and treated at dose level 1 are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 5
Participants
  Grade 2+ | 1
  Grade 3+ | 4
  Grade 4+ | 0

5. Secondary Outcome: Overall Response Rate (Phase II)
Description: The proportion of responses by 6 months will be estimated by the number of patients who achieve a response by 6 months divided by the total number of evaluable patients. The proportion of responses by 12 months will be estimated in a similar manner. Exact binomial 95% confidence intervals for the true success proportions will be calculated.
Time Frame: Up to 12 months
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Progression (Phase II)
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: The time from registration to the earliest date of documentation of disease progression, assessed up to 2 years
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Adverse Events, Graded According to the Grading Scale for Hematologic Adverse Events in CLL Studies (Phase II)
Description: The maximum grade for each type of adverse event, regardless of causality, will be recorded and reported for each patient, and frequency tables will be reviewed to determine adverse event patterns.
Time Frame: Up to 30 days after the last day of study treatment
Population: Trial terminated early with too few patients to analyze this endpoint.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected after each 28 day cycle of treatment for up to 4 cycles.
Description: Adverse Events were collected after each 28 day cycle of treatment for up to 4 cycles.
Arm/Group | Dose Level 1 (Lenalidomide in Combination With AT-101)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Lenalidomide in Combination With AT-101) (N=5)
Fatigue (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (Lenalidomide in Combination With AT-101) (N=5)
Anemia (Blood and lymphatic system disorders) | 5 (13)
Constipation (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (9)
Platelet count decreased (Investigations) | 5 (12)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT01003769/Prot_SAP_000.pdf